CLINICAL TRIAL: NCT01005693
Title: Impact of Frailty in Senior Cancer Patients: Feasibility and Value of Screening Tools and Geriatric Intervention and Predictive Value of a Screening Tool in Relation to Treatment Outcome
Brief Title: Screening Tools to Predict Treatment Outcome in Older Cancer Patients Who Are Undergoing Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: ZNA-2008-FOD-GER001; CDR0000658351 (Registry Identifier: PDQ (Physician Data Query)); EU-20985
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2010-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Mental Status and Dementia Tests; Restraint, Physical

INTERVENTIONS:
Other: questionnaire administration
Procedure: cognitive assessment
Procedure: examination
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Questionnaires that measure how well older patients think, learn, remember, and make judgments and carry out daily activities may improve the ability to plan treatment for patients with cancer.

PURPOSE: This clinical trial is studying testing for fitness to undergo chemotherapy to see how well it works in predicting treatment outcomes in older patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the feasibility of applying screening tools (Groningen Frailty Indicator [GFI] and G8) and their relationship to treatment outcome in older patients with cancer undergoing standard treatment versus geriatric interventions.
* To compare the screening tools (GFI and G8) with a comprehensive geriatric assessment (CGA).
* To evaluate the predictive value of the screening tool to undergo standard anticancer treatment in terms of toxicity.
* To identify patients that can benefit from a geriatric intervention in order to be able to undergo standard anticancer treatment.

OUTLINE: This is a multicenter study.

All patients complete screening questionnaires (GFI, G8, and the standardized CGA which consists of the ADL (Katz index) and IADL; the Timed Up and Go; the Cancer and Leukemia Group B adaptation of Charlson Co-morbidity; the Mini Nutritional Assessment; the RAND Social Support Survey Instrument; the Folstein Mini Mental State Examination; and the Geriatric Depression Scale) before the start of anticancer treatment, prior to each course of treatment, and after 1 month of treatment. Patients also undergo physical and cognitive performance measures by a trained member of the research team. Patients are assigned to a group based on fitness for treatment. They may be reassigned after each round of assessments.

* Group 1 (fit to undergo standard treatment): Patients undergo standard treatment.
* Group 2 (vulnerable): Patients receive specialized care and individualized treatment.
* Group 3 (frail): Patients receive palliative care and no anticancer chemotherapy or targeted agents.

Patients' medical history, vital signs, performance status, physical examination, and body weight are obtained and recorded. In patients receiving anticancer treatment, all adverse events are graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) and recorded and serious adverse events will be reported according to European Rules.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cancer

  * Undergoing out-patient care
  * Planning to undergo primary chemotherapeutic treatment or treatment with targeted agents for curative or palliative intent
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* Able to understand the Flemish language, give informed consent, and be followed at the investigational site
* Must be considered eligible for trial participation by the Investigator
* No severe known dementia
* No pre-existing major neurological or psychiatric problems
* No refusal of the standard anticancer strategy as defined by the service instruction book

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of applying screening tools (Groningen Frailty Indicator [GFI] and G8) in older patients with cancer
Comparison of the screening tools (GFI and G8) with a comprehensive geriatric assessment (CGA)
Predictive value of the screening tool to undergo standard anticancer treatment in terms of toxicity according to the NCI-CTC

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schrijvers, MD, PhD, Principal Investigator — Ziekenhuis Netwerk Antwerpen (ZNA)
Locations (4):
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Virga Jesse Hospital, Hasselt